CLINICAL TRIAL: NCT06036251
Title: COVID-19 Pandemic Induced Stress and Symptoms - Follow-up Study
Brief Title: COVID-19 Pandemic Induced Stress and Symptoms
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 23804; NCI-2023-06245 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Stress Reaction; Stress, Emotional; Stress; COVID-19 Pandemic
Keywords: Follow-up Study
MeSH Terms: conditions — Fractures, Stress; Stress, Psychological; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prior oncology participants: Oncology patients at University of California, San Francisco who participated in the previous study which evaluated the additional stressors imposed by COVID-19 (i.e., social isolation, loneliness) and ongoing general and disease specific stress on the symptom burden of cancer patients and survivors.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Self-reported quality of life (QOL) measures completed online

SUMMARY:
The previous survey of oncology patients at University of California, San Francisco in 2020-2021 found an alarmingly high symptom burden and high levels of stress and loneliness among respondents. This is a follow-up study with the same sample of oncology patients and survivors who participated in the previous study

DETAILED DESCRIPTION:
OBJECTIVES:

1. Evaluate for associations among general and disease-specific measures of stress and measures of social isolation and loneliness.
2. Evaluate for associations between general and disease-specific stress and common symptoms associated with cancer and its treatments.
3. Evaluate for associations between social isolation and loneliness and common symptoms associated with cancer and its treatments.
4. Evaluate for associations between social isolation and loneliness and health behaviors and quality of life (QOL) as compared to our last survey. as a baseline.
5. Evaluate for changes in stress, social isolation, loneliness and symptom burden between the two time points.

OUTLINE:

Patients will be asked to complete self-report questionnaires online. Questionnaires will take approximately 60 minutes to complete. and directed to take rest periods at 20 minute intervals. Participants will be given two weeks to complete the instruments.

ELIGIBILITY:
Inclusion Criteria:

* Current/Previous diagnosis of cancer
* Able to read, write, and understand English
* Able to complete the study questionnaires on line
* Able consent to participate.

Exclusion Criteria:

* Participants of our previous COVID survey study who opted out of future research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only previous patients and survivors who took part in our last COVID survey in 2020-2021 who agreed to be re-contacted for future research at University of California, San Francisco
Sampling Method: Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Correlation of scores on perceived stress scale (PSS) and social isolation scale (SIS) | 2 days
  Scores on the Perceived Stress Scale (PSS) from the previous study and this study, along with scores on the Social Isolation Scale (SIS) from the previous study, this study will be compared. The PSS is a 10-item questionnaire which asks participants about feelings and thoughts during the last month. Scores of each item ranging from 0 = "Never" to 4 = "Very Often" for a total score range of 0 to 40. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to 4 of the 10 positively stated items and scores are calculated by summing the total. Higher scores indicate higher degree of perceived stress. The Social Isolation Scale (SIS) is a measure used to assess an individual's tendency to isolate themselves from social situations. Scores on this scale are distributed with a mean of 15.0 and a standard deviation of 4.5.
Correlation of scores on the perceived stress scale (PSS) and loneliness scale | 2 days
  Scores on the Perceived Stress Scale (PSS) from the previous study and this study, along with scores on the University of California, Los Angeles (UCLA) Loneliness Scale from the previous study, and this study will be compared. The PSS is a 10-item questionnaire which asks participants about feelings and thoughts during the last month. Scores of each item ranging from 0 = "Never" to 4 = "Very Often" for a total score range of 0 to 40. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to 4 of the 10 positively stated items and scores are calculated by summing the total. Higher scores indicate higher degree of perceived stress. The 3-item UCLA loneliness scale is a 3-item scale used for measuring loneliness with scores ranging from 1='Hardly ever" to 3=Often. Scores are summed to generate a total score with higher scores indicating a higher degree of loneliness.
Correlation of scores on the perceived stress scale (PSS) and symptom severity scores | 2 days
  Scores on the PSS from the previous study and this study, along with scores on Memorial Symptom Assessment Scale (MSAS) from the previous study, and this study will be compared. The PSS is a 10-item questionnaire which asks participants about feelings and thoughts during the last month. Scores of each item ranging from 0 = "Never" to 4 = "Very Often" for a total score range of 0 to 40. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to 4 of the 10 positively stated items and scores are calculated by summing the total. Higher scores indicate higher degree of perceived stress. The MSAS is used to assess common physical symptoms experienced by persons with cancer. The values for severity and frequency measurements are 1='slight' or 'rarely' and 4= 'very severe'/'almost constantly' .Higher values indicate a greater number of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Miaskowski, RN,PhD,FAAN, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miaskowski C, Paul SM, Snowberg K, Abbott M, Borno HT, Chang SM, Chen LM, Cohen B, Cooper BA, Hammer MJ, Kenfield SA, Kober KM, Laffan A, Levine JD, Pozzar R, Rhoads K, Tsai KK, Van Blarigan EL, Van Loon K. Loneliness and symptom burden in oncology patients during the COVID-19 pandemic. Cancer. 2021 Sep 1;127(17):3246-3253. doi: 10.1002/cncr.33603. Epub 2021 Apr 27. PMID 33905528
- [Background] Miaskowski C, Paul SM, Snowberg K, Abbott M, Borno H, Chang S, Chen LM, Cohen B, Hammer MJ, Kenfield SA, Kober KM, Levine JD, Pozzar R, Rhoads KF, Van Blarigan EL, Van Loon K. Stress and Symptom Burden in Oncology Patients During the COVID-19 Pandemic. J Pain Symptom Manage. 2020 Nov;60(5):e25-e34. doi: 10.1016/j.jpainsymman.2020.08.037. Epub 2020 Sep 2. PMID 32889039
- [Background] Miaskowski C, Paul SM, Snowberg K, Abbott M, Borno H, Chang S, Chen LM, Cohen B, Cooper BA, Hammer MJ, Kenfield SA, Laffan A, Levine JD, Pozzar R, Tsai KK, Van Blarigan EL, Van Loon K. Oncology patients' perceptions of and experiences with COVID-19. Support Care Cancer. 2021 Apr;29(4):1941-1950. doi: 10.1007/s00520-020-05684-7. Epub 2020 Aug 18. PMID 32809060